CLINICAL TRIAL: NCT07036185
Title: An Open-Label, Multicenter, Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of KJ015 Injection (Subcutaneous Injection) in Patients With HER2-Expressing Solid Tumors
Brief Title: A Clinical Trail of KJ015 in Patients With HER2-Expressing Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Bao Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHBJ-KJ015-001
Record Dates: First submitted 2025-06-10; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Gastric/Gastroesophageal Junction Cancer; Breast Cancer; Colorectal Cancer; Non-small Cell Lung Cancer (NSCLC); Bile Duct Cancer; Head and Neck Squamous Cell Carcinoma
Keywords: KJ015; HER2; solid tumors
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Bile Duct Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Injections, Subcutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KJ015 Injection (Subcutaneous Injection) (Experimental): KJ015 is administered via subcutaneous injection.
  Interventions: Drug: KJ015 Injection (Subcutaneous Injection)

INTERVENTIONS:
Drug: KJ015 Injection (Subcutaneous Injection) — KJ015 is administered via subcutaneous injection, with the dosing frequency set at either Q3W.

SUMMARY:
This is an open-label, multicenter, Phase 1 study to evaluate the safety, tolerability, PK, and preliminary efficacy of KJ015 administered subcutaneously in participants with HER2-expressing solid tumors.

DETAILED DESCRIPTION:
This is an open-label, multicenter, Phase 1 study to evaluate the safety, tolerability, PK, and preliminary efficacy of KJ015 administered subcutaneously in participants with HER2-expressing solid tumors. The study will be conducted in 2 parts: the first part is the dose escalation part, and the second part is the Backfill part (as determined by the Sponsor). The dose escalation part will evaluate the safety and tolerability of KJ015 in participants with HER2-expressing locally advanced or metastatic solid tumors who have no standard therapy, are ineligible for surgical resection, or are not suitable for standard therapy or other approved therapies but have an inadequate clinical response. The Backfill part will further characterize the preliminary efficacy and safety of KJ015 in selected participants with solid tumors (including but not limited to G/GEJ, BC, CRC, BDC, HNSCC, NSCLC, etc.) at a minimum of two safe and tolerable dose levels, explore the relationship between the expression levels of HER2 protein and its mRNA and efficacy, as well as the HER 2 protein expression levels, transcription levels, and the correlation with efficacy in antitumor activity after KJ015 treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years (at time of free and informed consent).
2. Participants must have radiographically confirmed progressive disease (PD) during the last treatment prior to the first dose of enrollment.
3. Eastern Cooperative Oncology Group Performance Status (ECOG PS) Dose Escalation Part: ECOG performance status 0 to 1;Backfill Part: ECOG performance status0 to 2.
4. Participants must be have HER 2 positive or HER 2 expressing tumors determined by a certified local or central clinical laboratory or hospital
5. Organ function must meet the following criteria:

   i.Hemoglobin (Hb) ≥ 9.0 g/dL ii.Absolute neutrophil count (ANC) ≥ 1.0 × 109/L iii.Platelet count (PLT) ≥ 80 × 109/L v.Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN if no liver lesions (primary or metastatic); ALT and AST ≤ 5 × ULN if liver lesions are present vi.Creatinine clearance ≥ 30 mL/min vii.Activated partial thromboplastin time (APTT) and international normalized ratio (INR) ≤ 1.5 × ULN viii. Serum albumin ≥ 25 g/L (2.5 g/dL).
6. Expected survival ≥ 3 months.
7. Participants must be capable of and willing to comply with the visit and procedure requirements outlined in the protocol.

Exclusion Criteria:

1. Concurrent participation in another clinical study.
2. Received radiotherapy within 2 weeks prior to the first dose.
3. Underwent major surgery (excluding diagnostic surgery) within 4 weeks prior to the first dose or plan to undergo major surgery during the study. Underwent interventional or ablation surgery aimed at treating the tumor within 2 weeks before the first dose.
4. Prior allogeneic bone marrow transplant or prior solid organ transplant.
5. Received systemic corticosteroids or other immunosuppressive treatments within 2 weeks prior to the first dose.
6. Received an anthracycline cumulative dose of doxorubicin exceeding 500 mg/m2 or an equivalent dose of other anthracyclines prior to the first dose.
7. History of leptomeningeal carcinomatosis or carcinomatous meningitis.
8. Brain metastasis or spinal cord compression.
9. Uncontrolled or clinically significant cardiovascular or cerebrovascular disease.
10. History of a serious allergic reaction to the investigational product, an inactive ingredient in the investigational product, or other monoclonal antibody.
11. Women who are pregnant or breastfeeding as confirmed by pregnancy testing within 3 days prior to first dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-06-24 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation Part: Adverse Event collection and assessment | at least 21 days or up to 24 weeks
  Adverse Event collection and assessment will be done for all potentially treated subjects to assess the safety, tolerability, and determine the DLTs, maximum tolerated dose (MTD).
Dose Escalation Part: Backfill part recommended extension dose (RED) | at least 21 days or up to 24 weeks
  Backfill recommended extension dose
Backfill Part: Adverse Event | at least 21 days or up to 24 weeks
  Adverse Event collection and assessment will be done for all potentially treated subjects to assess the safety, tolerability.

SECONDARY OUTCOMES:
Immunogenicity | day 1, day 15, every 3 weeks
  Immunogenicity of KJ1015 (Anti-KJ015 antibody) in patients
Objective Response Rate (ORR) | at least 12 weeks
  ORR was defined as the patients with a best overall response of complete response (CR) or partial response (PR) based on local Investigator assessment as defined in RECIST 1.1.
Disease Control Rate (DCR) | at least 12 weeks
  DCR was defined as the patients with a best overall response of either CR, PR or stable disease (SD) .
Progression-Free Survival（PFS） | at least 12 weeks
  PFS was defined as the time from first dose of study treatment until the date of disease progression or death (by any cause in the absence of progression) regardless whether the patient withdrew from the assigned study treatment or received another anticancer prior to progression.
Overall Survival (OS) | at least 12 weeks
  OS was defined as the time from first day of study treatment until death due to any cause.
Maximum Observed Plasma Concentration (Cmax) | Pre-dose, 2-24, 48, 72, 96, 144-480 hours post-dose
  Maximum observed serum concentration of KJ015 following dosing (Cmax)
Terminal Half-life (t½) | Pre-dose, 2-24, 48, 72, 96, 144-480 hours post-dose
  Half-life of KJ015
Area under the serum concentration versustime curve (AUC) | Pre-dose, 2-24, 48, 72, 96, 144-480 hours post-dose
  Area under the serum concentration versustime curve (AUC) of KJ015
Apparent Volume of Distribution (Vz) | Pre-dose, 2-24, 48, 72, 96, 144-480 hours post-dose
  The PK (Vz) of KJ015
Clearance(CL) | Pre-dose, 2-24, 48, 72, 96, 144-480 hours post-dose
  Clearance(CL) is a measure of the ability of the body to clear KJ015

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No